CLINICAL TRIAL: NCT02542787
Title: A Phase II Proof of Concept (PoC), Double-Blind, Randomised, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of VSN16R for the Treatment of Spasticity in Subjects With Multiple Sclerosis
Brief Title: Study of VSN16R for the Treatment of Spasticity in Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canbex Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBX-001
Record Dates: First submitted 2015-09-04; First posted 2015-09-07 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Spasticity in People With Multiple Sclerosis
Keywords: MS; Spasticity; VSN16R
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental): VSN16R (Canbex name for molecule) oral capsules, 50mg-400mg daily or twice daily, total exposure 26 days
  Interventions: Drug: VSN16R
- Placebo (Placebo Comparator): Placebo capsules, 50mg-400mg daily or twice daily, total exposure 26 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: VSN16R — Small molecule
  Other Names: Not yet available
  Arms: Active
Other: Placebo — dummy tablet
  Arms: Placebo

SUMMARY:
Phase II a Proof of concept study in Multiple Sclerosis (MS) patients with spasticity.

DETAILED DESCRIPTION:
Single dose escalation followed by multiple fixed dose administrations to assess short term safety and to determine whether spasticity improves.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of MS
* Have an Expanded Disability Status Scale (EDSS) ≤ than 6.5 at screening.
* Spasticity due to MS of at least 3 months duration with minimum mean score of >/=2 mASH

Exclusion Criteria:

* Acute MS relapse requiring treatment with steroids within 30 days of screening.
* Initiation or discontinuation of MS disease modifying treatment (DMT) within 30 days of screening.
* Receiving medications that would potentially interfere with the actions of the study medication or outcome variables
* Significant renal and hepatic abnormalities
* Previous history of other significant medical disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale | 26 days

SECONDARY OUTCOMES:
Modified Ashworth Scale | 26 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr Rachel Farrell, Principal Investigator — University College London Hospitals
Locations (4):
- United Kingdom (4):
  - The Neuroscience Research Centre, The Walton Centre NHS Foundation Trust, Liverpool
  - The Royal London Hospital, London
  - The National Hospital for Neurology and Neurosurgery, London
  - Royal Hallamshire Hospital, Sheffield Teaching Hospital NHS Foundation Trust, Sheffield